CLINICAL TRIAL: NCT00421876
Title: GlObal Secondary Prevention strategiEs to Limit Event Recurrence After Myocardial Infarction. GOSPEL Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Care Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 60
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2007-01

CONDITIONS: Myocardial Infarction
Keywords: cardiac rehabilitation; lifestyle management; risk factor management; myocardial infarction; randomized trials
MeSH Terms: conditions — Myocardial Infarction

INTERVENTIONS:
Behavioral: multifactorial continued educational - behavioural programme

SUMMARY:
Cardiac rehabilitation programmes are a proven treatment for individuals with recent myocardial infarction, resulting in reduced morbidity and mortality compared to usual care. Unfortunately, following completion of a cardiac rehabilitation programme, risk factors and lifestyle behaviours may deteriorate. The GOSPEL study investigates the benefits of a programme of continued educational and behavioural intervention to achieve optimal long-term secondary prevention goals.

DETAILED DESCRIPTION:
Study partially sponsored by Società Prodotti Antibiotici

ELIGIBILITY:
Inclusion Criteria:

* Recent myocardial infarction (within 3 months after the index event)
* Standard rehabilitation program of 3-6 weeks performed
* Informed consent (obtained before any study specific procedure)

Exclusion Criteria:

* Age > 75 years
* Any condition that in the opinion of the investigator would jeopardize the evaluation of efficacy or be associated with poor adherence to the protocol;
* Presence of any non-cardiac disease (e.g. cancer) that is likely to significantly shorten life expectancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200
Dates: Start 2000-12; Study Completion 2005-12

PRIMARY OUTCOMES:
cardiovascular mortality
non fatal re-MI
angina requiring hospitalization
urgent revascularization procedures
hospitalization for heart failure
non fatal stroke

CONTACTS AND LOCATIONS:
Overall Officials: Pantaleo Giannuzzi, MD, Study Chair — Fondazione Maugeri - Veruno (NO)
Locations (74):
- Italy (73):
  - Ospedale San Donato, Arezzo, AR
  - Az Osp Giuseppe Moscati, Avellino, AV
  - Fondazione Salvatore Maugeri, Cassano delle Murge, BA
  - Ospedale Romano di Lombardia, Romano Lombardo, BG
  - Fondazione Salvatore Maugeri, Telese Terme, BN
  - Ospedale Bellaria, Bologna, BO
  - Presidio Gazzaniga, Gazzaniga, BS
  - Fondazione Salvatore Maugeri, Gussago, BS
  - Azienda Ospedaliera S Anna e S Sebastiano, Caserta, CE
  - Casa di Cura Villa Pini d'Abruzzo, Chieti, CH
  - Ospedale Umberto I, Bellano, Como
  - Ospedale Santa Marta, Rivolta d'Adda, CR
  - Ospedale Civile Minervini, Mormanno, CS
  - Ospedale Civile C Chidichino, Trebisacce, CS
  - Ospedale Ascoli Tomaselli, Catania, CT
  - Ospedale Cannizzarro, Catania, CT
  - Azienda Ospedaliera Mater Domini, Catanzaro, CZ
  - Az Ospedaliera-Universitaria Careggi, Florence, FI
  - Ospedale La Colletta, Arenzano, GE
  - Polo Ospedaliero Rapallo S Margherita, Rapallo, GE
  - ospedale Generale Provinciale, Gorizia, GO
  - Ospedale San Leopoldo, Merate, Lecco
  - Presidio Ospedaliero F Ferrari, Casarano, LE
  - Ospedale Civile Bassa Val di Cecina, Cecina, LI
  - Ospedale Civile Campo di marte, Lucca, LU
  - Presidio di Riabilitazione Multifunzionale, Bozzolo, MI
  - Casa di Cura Ambrosiana, Cesano Boscone, MI
  - Ospedale San Gerardo, Monza, MI
  - Presidio Ospedaliero di Passirana, Passirana - Rho, MI
  - Fondazione Salvatore Maugeri, Tradate, MI
  - Fondazione Salvatore Maugeri, Veruno, Novara
  - Ospedale Buccheri la Ferla Fatebenefratelli, Palermo, PA
  - Casa di Cura San Giacomo, Ponte dell'Olio, PC
  - Ospedale di Camposanpiero, Camposanpiero, PD
  - Predisio Ospedaliero Città di Castello, Città di Castello, PG
  - Nuovo Ospedale S Giovanni Battista, Foligno, PG
  - Ospedale Calai, Gualdo Tadino, PG
  - Azienda Ospedaliera di Perugia, Perugia, PG
  - Ex Ospedale Grocco, Perugia, PG
  - ospedale della Val di Nievole, Pescia, Point
  - Ospedale Civile, Sacile, Pordenone
  - Fondazione Salvatore Maugeri, Montescano, PV
  - Azienda Ospedaliera San Carlo, Potenza, PZ
  - Casa di Cura Villa Maria Cecilia, Cotignola, RA
  - Ospedale Infermi, Rimini, RA
  - Policlinico Madonna della Consolazione, Reggio Calabria, RC
  - Ospedale Sant'Anna, Castelnovo ne' Monti, RE
  - Ospedale Civile San Sebastiano, Correggio, RE
  - Ospedale E Morelli, Sondalo, SO
  - Ospedale SS Annunziata, Taranto, TA
  - Ospedale di ALA, Ala, TN
  - Ospedale Provinciale S Pancrazio, Arco, TN
  - Presidio Ospedaliero, Montebelluna, TV
  - Ospedale Civile, Mirano, VE
  - Ospedale Civile, San Donà di Piave, VE
  - Ospedale Beauregard, Aosta
  - Ospedali Riuniti, Bergamo
  - Casa di Cura Villa Aprica, Como
  - Casa di Cura Pineta del Carso, Duino-Aurisina
  - Presidio Ospedalier S Giovanni, Mezzolombardo
  - Fondazione Don Gnocchi, Milan
  - Istituti Clinici Perfezionamento, Milan
  - Ospedale S Luca-Centro Auxologico, Milan
  - Pio Albergo Trivulzio, Milan
  - Azienda Ospedaliera Vincenzo Monaldi, Napoli
  - Policlinico Universitario Federico II, Napoli
  - Fondazione Salvatore maugeri, Pavia
  - Ospedale Forlanini, Roma
  - Ospedale Santo Spirito, Roma
  - Villa Betania, Roma
  - Ospedale Evangelico Valdese, Torino
  - Ospedale Mauriziano, Torino
  - ospedale Civile S Bortolo, Vicenza
- Cardiocentro Ticino, Lugano, Switzerland

REFERENCES:
- [Background] Giannuzzi P, Temporelli PL, Maggioni AP, Ceci V, Chieffo C, Gattone M, Griffo R, Marchioli R, Schweiger C, Tavazzi L, Urbinati S, Valagussa F; GOSPEL. GlObal Secondary Prevention strategiEs to Limit event recurrence after myocardial infarction: the GOSPEL study. A trial from the Italian Cardiac Rehabilitation Network: rationale and design. Eur J Cardiovasc Prev Rehabil. 2005 Dec;12(6):555-61. doi: 10.1097/01.hjr.0000186623.60486.26. PMID 16319545
- [Result] Giannuzzi P, Temporelli PL, Marchioli R, Maggioni AP, Balestroni G, Ceci V, Chieffo C, Gattone M, Griffo R, Schweiger C, Tavazzi L, Urbinati S, Valagussa F, Vanuzzo D; GOSPEL Investigators. Global secondary prevention strategies to limit event recurrence after myocardial infarction: results of the GOSPEL study, a multicenter, randomized controlled trial from the Italian Cardiac Rehabilitation Network. Arch Intern Med. 2008 Nov 10;168(20):2194-204. doi: 10.1001/archinte.168.20.2194. PMID 19001195